CLINICAL TRIAL: NCT02159872
Title: A Phase II Study of Omacetaxine (OM) in Patients With Intermediate-1 and Higher Risk Myelodysplastic Syndrome (MDS) Post Hypomethylating Agent (HMA) Failure
Brief Title: Omacetaxine in Patients With Intermediate-1 and Higher Risk Myelodysplastic Syndrome (MDS) Post Hypomethylating Agent (HMA) Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0870; NCI-2014-01483 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic Syndrome; MDS; Omacetaxine; Synribo; Homoharringtonine
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omacetaxine (Experimental): Omacetaxine 1.25 mg/m2 subcutaneously every 12 hours on Days 1-3 of every 28-day study cycle. Participant may continue taking the study drug for up to 24 cycles of treatment.
  Interventions: Drug: Omacetaxine

INTERVENTIONS:
Drug: Omacetaxine — 1.25 mg/m2 subcutaneously every 12 hours on Days 1-3 of every 28-day study cycle.
  Other Names: Synribo; Homoharringtonine

SUMMARY:
The goal of this clinical research study is learn if omacetaxine can help to control myelodysplastic syndrome (MDS). The safety of this drug will also be studied.

This is an investigational study. Omacetaxine is FDA approved and commercially available for the treatment of chronic myelogenous leukemia (CML). It is investigational to use omacetaxine in patients with MDS. The study doctor can explain how the study drug is designed to work.

Up to 80 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

Each cycle will be 4-7 weeks, depending on how well the disease responds to the study drug.

If you are found to be eligible to take part in this study, you will receive omacetaxine as an injection under your skin 2 times each day, about 12 hours apart, on Days 1-3 of every 28-day study cycle.

You will receive instructions on how to give these injections to yourself. You will be given a Research Drug Diary to record the drug you take each day. You must bring the Research Drug Diary and any unused drug with you to each study visit. You will also be told how to properly store the drugs.

Depending on how the disease responds to the study drugs, the number of days you receive your injections may stay the same, increase, or decrease. Your doctor will discuss this with you.

During Cycle 1, if the doctor thinks it is needed, you will be given hydroxyurea by mouth to decrease the risk of side effects. You may ask the study staff for information about how the drug is given and its risks.

Study Visits:

At the beginning of every cycle, you will have a physical exam before your dose of study drug.

Every week (+/- 2 days), blood (about 2-3 teaspoons) will be drawn for routine tests. If the disease appears to get better, this blood will only be drawn every 2-4 weeks while you are still receiving the study drugs.

If you live far from the clinic, this blood can be drawn at a clinic close to your home, and the results will be reported to the study doctor.

If the study doctor thinks it is needed, you may have an additional bone marrow aspirate at any time during the study to check the status of the disease and for cytogenetic testing.

Length of Study:

You may continue taking the study drug for up to 24 cycles of treatment. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Follow-Up:

You will have follow-up visits at the clinic every 3-6 months for up to 5 years after you stop taking the study drug. You will be asked about your health and any new drugs you may be taking. If you cannot come to the clinic, you will be called by the study staff and asked about your health. These calls should last about 5-10 minutes.

Every 4-8 weeks after your last dose of study drug, blood (about 2-3 teaspoons) will be drawn for routine tests.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. Diagnosis of MDS confirmed within 10 weeks prior to study entry according to WHO criteria. Patients are either not eligible for or choose not to proceed with a stem cell transplant.
3. MDS classified as follows: RAEB-1 (5%-9% BM blasts); RAEB-2 (10%-19% BM Blasts); CMML (5%-19% BM blasts); RAEB-t (20%-29% BM blasts) AND/OR by IPSS: intermediate-1 and high risk patients.
4. No response, progression, or relapse (according to 2006 IWG criteria) following at least 4 cycles of either azacitidine or decitabine, which were completed within the last 2 years - AND/OR - intolerance to azacitidine or decitabine defined as drug-related >/= grade 3 hepatic or renal toxicity leading to treatment discontinuation during the preceding 2 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of </= 2.
6. Willing to adhere to and comply with all prohibitions and restrictions specified in the protocol.
7. Patient (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.)

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
2. Active infection not adequately responding to appropriate antibiotics (i.e. ongoing temperatures of >/= 38 degree Celsius).
3. Total bilirubin >/= 1.5 mg/dL and not related to hemolysis or Gilbert's disease. Patients with total bilirubin >/= 1.5 mg/dL to 3 mg/dL are eligible if at least 75% of the bilirubin is indirect.
4. Alanine transaminase (ALT/SGPT) or aspartate transaminase (AST/SGOT) >/= 2.5 x the upper limit of normal.
5. Serum creatinine > 1.5 mg/dL.
6. Female patients who are pregnant or lactating.
7. Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study.
8. Female patients with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta HCG) pregnancy test at screening.
9. Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy.
10. Prior hydroxyurea for control of leukocytosis or use of hematopoietic growth factors (eg, G-CSF, GM-CSF, procrit, aranesp, thrombopoietins) is allowed at any time prior to or during study if considered to be in the best interest of the patient.
11. Psychiatric illness or social situation that would limit the patient's ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2015 to September 2018
Period: Overall Study
Arm/Group | Omacetaxine
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Omacetaxine
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 43
Age, Continuous [Median (Full Range); unit: years] | 75.5 [60 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 42
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time from treatment start to the time of death. Overall survival continuously monitored using the Bayesian method.
Time Frame: Up to 2.5 Years
Measure: Median (Full Range); unit: Months
Arm/Group | Omacetaxine
Number analyzed (Participants) | 48
Months | 7.5 [0.1 to 30]

2. Primary Outcome: Number of Participants With a Response
Description: Response is Complete Response (CR) + Partial Response (PR) + Hematologic Improvement (HI). CR is the normalization of the peripheral blood and bone marrow with </= 5% bone marrow blasts, a peripheral blood granulocyte count >/= (1.0x10^9/L, and a platelet count >/= 100x10^9/L). PR is the same as CR except for the presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment. HI meets all of the criteria for CR except for platelet recovery to >/=100x10^9L.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Omacetaxine
Number analyzed (Participants) | 48
Participants | 16

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Omacetaxine
All-Cause Mortality (participants affected / at risk) | 15/48
Serious Adverse Events (participants affected / at risk) | 30/48
Other Adverse Events (participants affected / at risk) | 23/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine (N=48)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Bacteremia Infection (Infections and infestations) | 1 (1)
Cardiac Ischemia (Cardiac disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Graft Versus Host Disease (General disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Left Shoulder Pain (General disorders) | 1 (1)
Oral Mucositis (Gastrointestinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nausea & Vomiting (Gastrointestinal disorders) | 1 (1)
Neoplasms benign, Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Arm Cellulitis (Infections and infestations) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Subaracnoid hemorrhage (Nervous system disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epigastric Pain (Gastrointestinal disorders) | 1 (1)
Right Cervical Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Gingival Infiltration (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fever, Flu Shot Reaction (Immune system disorders) | 1 (2)
Hypotension (Vascular disorders) | 2 (2)
RSV Pneumonia (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 2 (2)
Spasticity (Severe Muscle Spasm) (Musculoskeletal and connective tissue disorders) | 2 (2)
Multi-Organ Failure (General disorders) | 1 (1)
Lung Infection (Infections and infestations) | 3 (3)
Upper Gastrointestianl Hemorrhage (Gastrointestinal disorders) | 2 (3)
Fever (General disorders) | 5 (5)
Death (General disorders) | 7 (7)
Pneumonia (Infections and infestations) | 6 (7)
Neutropenic Fever (Blood and lymphatic system disorders) | 8 (13)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine (N=48)
Hemorrhage (General disorders) | 3 (3)
Forgetfulness (Nervous system disorders) | 4 (4)
Mouth Sores (Gastrointestinal disorders) | 4 (4)
Neutropenic Fever (Blood and lymphatic system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 5 (5)
Edema (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Infection (Infections and infestations) | 12 (12)
Nausea/Vomiting (Gastrointestinal disorders) | 20 (20)
Fatigue (General disorders) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT02159872/Prot_SAP_000.pdf